CLINICAL TRIAL: NCT04279080
Title: Low Anterior Resection Syndrome (LARS) in Ovarian Cancer Patients - a Multi-centre Comparative Analysis.
Brief Title: LARS in Ovarian Cancer Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Felix Harpain, Principle Investigator, M.D., Medical University of Vienna
Other Study IDs: 1201/2018
Record Dates: First submitted 2020-02-16; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: rectal cancer patients
  Interventions: Other: low anterior resection syndrome evaluation
- 2: ovarian cancer patients
  Interventions: Other: low anterior resection syndrome evaluation

INTERVENTIONS:
Other: low anterior resection syndrome evaluation — evaluation of postoperative functional bowel outcome

SUMMARY:
Background:

Low anterior resection syndrome (LARS) is a common functional disorder after low anterior resection impacting quality of life. Data on LARS derives nearly exclusively from rectal cancer studies. Therefore, the study was designed to assess LARS in advanced epithelial ovarian cancer (EOC) patients, who underwent rectal resection and to compare it with a female rectal cancer cohort.

Methods:

A cross-sectional multi-centre analysis was performed for female patients suffering from either rectal or EOC who received a low anterior resection as part of their therapy regimen. None of the patients received pre- or postoperative radiotherapy. LARS was defined by using the validated LARS score and its severity was divided into "no", "minor" and "major LARS".

ELIGIBILITY:
Inclusion Criteria:

* low anterior resection because of ovarian or rectal cancer

Exclusion Criteria:

* neoadjuvant or adjuvant radiotherapy

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cross-sectional multi-centre analysis was performed for female patients suffering from either rectal or EOC who received a low anterior resection as part of their therapy regimen.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
functional bowel outcome after low anterior resection | 1 year
  low anterior resection syndrome score, questionnaire via telephone call or personal contact